CLINICAL TRIAL: NCT04955990
Title: An International, Non-Drug Interventional, Real-world Cohort of PAH Patients Newly Initiating PAH Therapy With Guideline-directed Assessments of Disease Severity
Brief Title: A Study of Real-world Cohort of Pulmonary Arterial Hypertension (PAH) Participants
Acronym: CARE PAH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study.
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109007; 67896062PAH4005 (Other: Actelion)
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with PAH (Experimental): Participants with pulmonary arterial hypertension (PAH) who newly initiate any PAH therapy(ies) at the index date (date when a participant starts the first new PAH therapy after baseline assessments) in a routine clinical setting, either as first-line therapy, as replacement therapies, as concomitant with other PAH therapies, or have already been receiving macitentan 10 milligrams (mg) for at least 3 months prior to the index date. The primary data source for this study will be the medical records of each participant.
  Interventions: Other: PAH Therapies

INTERVENTIONS:
Other: PAH Therapies — No Drug will be administered as part of this study. Real world data will be collected in participants who newly initiate PAH therapies in routine clinical setting or have already been receiving macitentan 10 mg for at least 3 months prior to the index date.

SUMMARY:
This study is designed to describe pulmonary arterial hypertension (PAH) participants in terms of their clinical characteristics, therapies used, disease progression, and outcomes (example, death, hospitalization, risk category for predicted mortality risk, and patient-reported outcomes [PROs]) in real-world clinical practice. This study will collect high-quality real-world data that may be used as a stand-alone dataset or in combination with other studies to address relevant research questions (example, serve as an external control dataset to another study) to support development and access to PAH therapies, as well as to contribute to the knowledge base of PAH through publications.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary arterial hypertension (PAH) in any PAH subtype
* PAH diagnosis confirmed by hemodynamic evaluation at rest at any time prior to or at the index date fulfilling all of the criteria below: a) Mean pulmonary artery pressure greater than (>) 20 millimeters of mercury (mm Hg), and b) Pulmonary artery wedge pressure or left ventricular end diastolic pressure less than or equal to (<=) 15 mm Hg, and c) Pulmonary vascular resistance greater than or equal to (>=) 3 Wood Units (that is, >= 240 dynes seconds per centimeters penta [dyn∙sec/cm^5])
* Participant satisfies either a or b: a) Newly initiating 1 or more PAH therapy(ies) (as monotherapy or add-on therapy) at index date. These newly initiated PAH therapies should not have been used within 3 months of the index date; b) Taking macitentan 10 milligrams (mg) therapy (as monotherapy or in combination) with no changes in PAH therapy for within 3 months prior to the index date
* All mandated assessments must be performed and recorded at the baseline visit before the initiation of the new PAH therapy at the index date or enrollment in the study.
* For the pulmonary arterial hypertension-symptoms and impact (PAH-SYMPACT) substudy only: Participants initiating any endothelin receptor antagonist (ERA) or phosphodiesterase-5 inhibitor therapies at index date or at therapy change must provide consent to enroll in the optional PAH-SYMPACT substudy. Refusal to give consent for the optional PAH-SYMPACT substudy will not exclude a participant from participation in the main study

Exclusion Criteria:

* Participants enrolled in any interventional clinical trial with an investigational therapy in the 3-month period prior to index date
* Currently enrolled in an observational study sponsored or managed by a Janssen company
* Presence of moderate or severe obstructive lung disease (forced expiratory volume in 1 second [FEV1] / forced vital capacity [FVC] <70%; and FEV1 <60% of predicted after bronchodilator administration) in participants with a known or suspected history of significant lung disease, as documented by a spirometry test performed within 1 year prior to screening
* Presence of moderate or severe restrictive lung disease (for example, total lung capacity or FVC <60 percent [%] of normal predicted value) in participants with a known or suspected history of significant lung disease, as documented by a spirometry test performed within 1 year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Time to all Cause Death | Up to 6 years
  Time to all cause death will be reported. All-cause death defined as deaths due to any cause.
Time to Death due to Pulmonary Arterial Hypertension (PAH) or First Hospitalization due to PAH | Up to 6 years
  Time to death due to PAH or first hospitalization due to PAH will be reported.

SECONDARY OUTCOMES:
Time to Death due to PAH | Up to 6 years
  Time to death due to PAH will be reported.
Time to First all-cause Hospitalization | Up to 6 years
  Time to first all-cause hospitalization will be reported.
Time to First Morbidity/Mortality Event | Up to 6 years
  Time to first morbidity/mortality event will be reported. All-cause death, non-planned hospitalization due to PAH (including for worsening of PAH, atrial septostomy, lung transplantation with or without heart transplantation, or initiation of parenteral prostacyclins), PAH-related disease progression, defined as (both criteria must be satisfied): At least 15 percent (%) decrease in 6-minute walking distance (6MWD) from baseline or therapy change visit, and initiation of additional PAH therapy or worsening of World Health Organization (WHO) functional class (FC) will be collected for morbidity/mortality events assessment.
Time to Clinical Worsening | Up to 6 years
  Time to clinical worsening will be reported. All-cause death, non-planned hospitalization due to PAH (including for worsening of PAH, atrial septostomy, lung transplantation with or without heart transplantation, or initiation of parenteral prostacyclins), PAH-related deterioration identified by at least 1 criterion: worsening of WHO FC, deterioration by at least 15% in exercise capacity, as measured by the 6MWD, any signs or symptoms of right-sided heart failure will be collected for clinical worsening assessment.
Medical Resource Utilization | Up to 6 years
  Number per year of all-cause and PAH-related hospitalizations; number per year of in-patient hospital days for all causes and PAH-related causes; number per year of emergency room visits for all causes and for PAH-related causes that do not result in hospital admittance will be collected for assessment of medical resource utilization.
Change from Baseline in 6-minute Walk Distance (6MWD) | Baseline up to 6 years
  Change from baseline in 6MWD according to non-invasive criteria will be assessed as per the low (greater than [>] 440 meters [m]), intermediate (165-440m), and high-risk category (less than [<] 165m).
Change from Baseline in World Health Organization (WHO) Functional Class (FC) | Baseline up to 6 years
  Change from baseline in WHO FC according to non-invasive criteria will be assessed as per the low (I, II), intermediate (III), and high-risk category (IV).
Change from Baseline in N-terminal-pro-hormone Brain Natriuretic Peptide (NT-proBNP) | Baseline up to 6 years
  Change from baseline in NT-proBNP according to non-invasive criteria will be assessed as per the low (<300 nanogram per liters [ng/l]), intermediate (300-1400ng/l), and high-risk category (>1400 ng/l).
Time to Worsening in WHO FC | Up to 6 months
  Time to worsening in WHO FC will be reported.
Change from Baseline in the Number of low-risk Noninvasive Criteria Based on WHO FC, 6MWD, and NT-proBNP | Baseline up to 6 years
  Change from baseline in the number of low-risk noninvasive criteria based on WHO FC, 6MWD, and NT-proBNP will be reported.
Time to all-cause Death Based on the Number of low-risk Noninvasive criteria Based on WHO FC, 6MWD, and NT-proBNP | Up to 6 years
  Time to all-cause death based on the number of low-risk noninvasive criteria based on WHO FC, 6MWD, and NT-proBNP will be reported.
Change from Baseline in Number of Participants Within Each Overall Risk Category (Low, Intermediate, or High) According to the Noninvasive Criteria | Baseline up to 6 years
  Change from baseline in number of participants within each overall risk category (low, intermediate, or high) according to low-risk non-invasive criteria will be assessed as per the following parameters: WHO FC- low (I, II), intermediate (III), and high-risk category (IV); 6MWD- low (> 440m), intermediate (165-440m), and high-risk category (< 165m), and <165m; and NT-proBNP- low (<300ng/l), intermediate (300-1400ng/l), and high-risk category (>1400 ng/l).
Change from Baseline in Number of Participants Within Each Overall Risk Category (low, Intermediate, or High) According to Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) Lite 1 Variables | Baseline up to 6 years
  Change from baseline in number of participants within each overall risk category (low, Intermediate, or High) according to REVEAL Lite 1 Variables will be reported. The REVEAL Lite 1 variables risk calculator determines the risk status, and the scores (ranges from 0 to 19) can be defined as: low risk as a score of less than or equal to (<=) 6, intermediate risk as a score of 7 or 8, and high risk as a score of greater than or equal to (>=) 9 for the survival rates.
Change from Baseline in Number of Participants Within Each Overall Risk Category (low, Intermediate, or High) According to REVEAL Lite 2 Variables | Baseline up to 6 years
  Change from baseline in number of participants within each overall risk category (low, Intermediate, or High) according to REVEAL Lite 2 Variables will be reported. The REVEAL Lite 2 variables risk calculator determines the risk status, and the scores (ranges from 1 to 14) can be defined as: low risk as a score of <= 5, intermediate risk as a score of 6 or 7, and high risk as a score of >= 8 for the survival rates.
Time to all-cause Death Based on the Risk Category Determined by the Noninvasive Criteria | Up to 6 years
  Time to all-cause death based on the risk category determined by the noninvasive criteria will be reported.
Time to all-cause Death Based on the Risk Category Determined by the REVEAL Lite 1 | Up to 6 years
  Time to all-cause death based on the risk category determined by the REVEAL Lite 1 will be reported.
Time to all-cause Death Based on the Risk Category Determined by the REVEAL Lite 2 | Up to 6 years
  Time to all-cause death based on the risk category determined by the REVEAL Lite 2 will be reported.
Risk Assessment Strategies for Clinical Worsening or Death | Up to 6 years
  The assessment of risk category for clinical worsening and death will be assessed by the following 3 risk assessment strategies: number of low-risk noninvasive criteria based on WHO FC, 6MWD, and NT-proBNP.
Change from Baseline in Health-related Quality of Life (HRQoL) as Measured by Symptoms and Impact Questionnaire for Use in Clinical Practice (SYMPACT-CP) Questionnaire | Baseline up to 6 years
  A modified version of the PAH-SYMPACT for Use in Clinical Practice (SYMPACT-CP), has been created for use in routine clinical practice, as an assessment to support symptom monitoring and guide treatment decisions by healthcare providers. In the SYMPACT-CP, the 24-hour recall period for the oxygen use item and the 11 symptoms items have been modified to a 1-week recall period. The SYMPACT-CP also includes 11 impact items (with a 1-week recall period). This modification was made with the intention of administering the questionnaire at a single timepoint.
Change from Baseline in Health Related Quality of Life Assessed by European Quality of Life (EuroQoL) Group, 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) | Baseline up to 6 years
  The EQ-5D-5L is an instrument to measure health-related quality of life consisting of a descriptive system and visual analogue scale (VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of perceived problems (1 indicating no problem, 2 indicating slight problems, 3 indicating moderate problems, 4 indicating severe problems, 5 indicating extreme problems). Participant selects an answer for each of 5 dimensions considering the response that best matches his or her health "today". The responses to the 5 dimensions are used to compute a single score ranging from 0 (worst health state) to 100 (better health state) representing the general health status of the individual.
Change from Baseline in Health-Related Quality of life Status as Assessed by 36-item Short-Form Health Survey (SF-36) v2 Acute Questionnaire | Baseline up to 6 years
  The SF-36 v2 acute questionnaire is a 36-item short form survey used to assess the participant's quality of life. In the SF-36 v2 Acute Questionnaire, participants are instructed to rate their health and capacity to perform activities of daily living in eight domains including physical functioning, physical role limitations, bodily pain, general health, vitality, social functioning, emotional role limitations, and mental health during the last week. The scores range from 0 (lowest or worst possible level of functioning) to 100 (highest or best possible level of functioning).
Change from Baseline in PAH-specific Medication Adherence as Assessed by Morisky Medication Adherence Scale-8 (MMAS-8) Score | Baseline up to 6 years
  The MMAS-8 is commonly used in standard clinical practice and a validated measure of treatment adherence. The MMAS-8 includes 8 questions assessing the extent of adherence or nonadherence and reasons for non-adherence.
Change from Baseline in Medication Adherence Questions of each Prescribed PAH Therapy Class | Baseline up to 6 years
  Change from baseline in medication adherence questions of each prescribed PAH therapy class will be reported.
Change from Baseline in PAH-specific Medication Adherence as Assessed by Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire | Baseline up to 6 years
  The PAH-SYMPACT questionnaire, applicable only for participants who enrolled in the PAH-SYMPACT substudy, is a PRO instrument and composed of 2 parts: the symptoms part and the Impacts part. There is no total symptom score; the 2 domains are: cardiopulmonary symptoms and cardiovascular symptoms. The Impacts part has 2 domains: Physical Impacts Domain and Cognitive/Emotional Impacts Domain which contain 7 and 4 items, respectively. Each item has 5-point Likert response scale (0=not at all, 1=mild, 2=moderate, 3=severe, and 4=very severe). The mean individual weekly symptom item scores are aggregated by domain, with the sum then being divided by the number of symptom items in the respective domain. This leads to the average weekly domain score ranging from 0-4 for each participant with higher scores indicating greater symptom severity or worse impact.
Change from Baseline in Patient Global Assessment of Disease Severity (PGA-S) of PAH | Baseline up to 6 years
  Change from baseline in PGA-S of PAH will be reported. It includes severity of PAH symptoms, such as, none, mild, moderate, severe and very severe.
PAH Symptoms and Impact using SYMPACT-CP Questionnaire | Baseline up to 6 years
  PAH symptoms and impact using SYMPACT-CP questionnaire will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (54):
- United States (15):
  - Bay Area Cardiology Associates, P.A. - Brandon Office, Brandon, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University Of Iowa - Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Cinncinnati Physicans- UC Health Physicnas Office, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
- Instituto Cardiovascular de Rosario, Rosario, Argentina
- Brazil (4):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre Victoria Hospital, London, Ontario
- China (5):
  - Beijing Anzhen Hospital, Beijing
  - Beijing Fuwai Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Shanghai Pulmonary Hospital, Shanghai
- Universitatsklinikum Bonn, Bonn, Germany
- Italy (3):
  - Ospedale S.Giuseppe, Gruppo MultiMedica, Milan
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Universita degli Studi di Roma 'La Sapienza' - Umberto I Policlinico di Roma, Rome
- National Hospital Organization Okayama Medical Center, Okayama, Japan
- National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (3):
  - Vrije Universiteit Amsterdam (VU), Amsterdam
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- Poland (2):
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
- CardioPulmonary Research, PSC, Guaynabo, Puerto Rico
- National Heart Centre (NHC) Singapore, Singapore, Singapore
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (3):
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Univ. Marques de Valdecilla, Santander
- Sahlgrenska Universitetsjukhuset, Gothenburg, Sweden
- United Kingdom (5):
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Papworth Hospital, Cambridge University, Papworth Everard
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency